CLINICAL TRIAL: NCT05750433
Title: PHAGE 3: Determination of Phage and Probiotic Synergistic Effects on Gastrointestinal Health
Brief Title: Phage 3Determination of Phage/Probiotic Synergistic Effects on Gastrointestinal Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Archer Daniels Midland Company (Unknown)
Responsible Party: Principal Investigator, Tiffany Weir, Associate Professor of Nutrition and Food Science, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1676
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Gastrointestinal Dysfunction
Keywords: PreforPro; Probiotics; Bacillus subtilis; Prebiotics; Gut health; Gut microbiota; Synergistic effects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, study personnel, and outcomes assessor are all blinded to treatment group. Blinding was completed by an independent individual that was not associated with the study or the sponsors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PreforPro+B. subtilis DE111 probiotics (Experimental): PreforPro is a prebiotic which is a bacteriophage-based product. This prebiotic was used in combination with Bacillus subtilis probiotics.
  Interventions: Dietary Supplement: PreforPro+B. subtilis DE111 probiotics
- Placebo(maltodextrin) (Placebo Comparator): Maltodextrin was used as a placebo.
  Interventions: Dietary Supplement: Placebo
- B. subtilis DE111 alone (Active Comparator): Bacillus subtilis probiotics was used in this arm alone to compare with the experimental arm.
  Interventions: Dietary Supplement: B. subtilis DE111

INTERVENTIONS:
Dietary Supplement: PreforPro+B. subtilis DE111 probiotics — PreforPro is bacteriophage-based product which was used in combination with Bacillus subtilis probiotics.
  Arms: PreforPro+B. subtilis DE111 probiotics
Dietary Supplement: Placebo — Maltodextrin is rice based powder which was used as placebo.
  Arms: Placebo(maltodextrin)
Dietary Supplement: B. subtilis DE111 — Bacillus subtilis probiotics.
  Arms: B. subtilis DE111 alone

SUMMARY:
The goal of this double blinded clinical trial is to determine whether consumption of the PreforPro product, when co-consumed with Bacillus subtilis DE111 probiotic, synergistically improves bowel regularity, perceived physical symptoms of gastrointestinal distress and other aspects of gastrointestinal health over probiotic use alone. Therefore, the primary goal of this study is to see if PreforPro consumption concurrent with B. subtilis DE111 usage improves probiotic activity. The secondary goal of this study is to assess non-gastrointestinal physiologic parameters to determine whether consumption of PreforPro combined with the probiotic offers any additional health benefits (ie. reduced inflammation, improved gut microbiota profiles) beyond those of consuming a probiotic alone.

Participants will be asked to track daily bowel movements for 7 days prior to beginning capsule consumption and record their diet for a total 3 of days (two weekdays and one weekend day). They will then be asked to consume the provided capsules daily for a period of 45 days. Researchers will compare three parallel arms; (1) PreforPro+B. subtilis DE111 probiotic, (2) B. subtilis DE111 alone, or (3) a maltodextrin placebo to establish their impact on gastrointestinal symptoms and other indicators of health.

DETAILED DESCRIPTION:
This is a continuation of previous intervention studies exploring the impacts of a bacteriophage formulation, PreforPro, on gastrointestinal health. The purpose of this study is to determine if the PreforPro product acts synergistically with a spore-based probiotic to influence bowel habits, perceptions of gastrointestinal symptoms, microbiota composition and inflammatory and immune parameters. The proposed study will also explore a longer intervention duration than the previous studies. A secondary outcome will include measuring plasma lipids, as the proposed probiotics (B. subtilis DE111) was shown to improve total and LDL cholesterol levels in our previous study. Bacteriophages may directly influence the microbiota and intestinal environment by selectively infecting host species- in this case E. coli. Additionally, they may have indirect effects as infection of target species can open up ecological niches and/or result in assimilation of released nutrients by other commensal organisms. These phages are generally regarded as safe for human consumption and specifically infecting several strains of E. coli, including enterohemorrhagic strains and Shiga-toxin producing strains. The removal of these E. coli alters the gut environment to allow growth of more favorable bacteria. We have previously shown that PreforPro is both safe and tolerable in a human population and does not broadly disrupt the gut microbiota as would be seen with antibiotic treatment. It did not improve the survival of Bifidobacterium lactis probiotic, but did appear to amplify some of its impacts on perceived functional gastrointestinal health.

A phone screening will be conducted of all interested individuals to evaluate their eligibility. Those meeting the initial eligibility criteria will be scheduled for a clinic visit to obtain informed consent and to confirm eligibility. Consent will be obtained at the Colorado State University Food and Nutrition Clinical Research Lab (FNCRL) by a screening questionnaire and interview/assessment by the clinical coordinator. After securing consent, eligibility will be confirmed by taking anthropometric measures and participants falling within the BMI range will randomly be assigned to 1 of 3 treatment groups: (1) PreforPro+B. subtilis DE111 probiotic, (2) B. subtilis DE111 alone, or (3) maltodextrin placebo.

Visit 1 (baseline): Eligible individuals will be asked to visit the clinic at visit 1 (baseline) to provide consent and confirm eligibility, undergo sample collections (blood and stool) and analysis procedures (weight/height, hip:waist ratio, gastrointestinal symptoms/ quality of life questionnaires) and receive their stool collection container, a stool log and 3-day diet log. Participants will be schedule for their drop off visit, in which they will return to the clinic 7 days after their first visit (Visit 2, Day 0) to return their stool sample, stool log and 3-day diet record. In return, they will be provided with another stool collection kit, their treatment capsules, another stool log and 3-day diet log. At the end of the 45-day treatment period (Visit 3-Final), final blood and stool samples will be collected as well as additional analyses (such as GI questionnaires, stool logs and 3-day diet record). This means that participants will undergo screening (by phone) and make a total of three (3) visits to the clinic during the study (baseline, Day 0, Final). All blood samples will be collected at Colorado State University by trained personnel. Fecal sample collection will be performed by the study participant with collection materials provided by Colorado State University.

ELIGIBILITY:
Inclusion Criteria:

* Equal numbers of healthy male and female volunteers between 18-75 years old with BMI scores of 18.5 to 34.9.

Exclusion Criteria:

* Individuals less than 18years of age or greater than 75years of age.
* If an individual's BMI is outside of 18.5-34.9.
* History of taking antibiotics and/or probiotics/prebiotics supplementation within 2months of starting antibiotics.
* If individual is on any medications and dietary supplements that would influence the endpoints of the study, such as statins, metformin, NSAIDs and MAO inhibitors.
* If individuals with diagnosis with cancer, liver or kidney disease, gastrointestinal diseases and metabolic disorders.
* Pregnant and breastfeeding women.
* Additionally inclusion and exclusion in the study will be determined case by case based on self reported alcohol and supplement use.
* If individual is unable to adhere to study protocol such as consuming capsules for a total 45days, providing stool or blood samples and attending scheduled clinic visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-23 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Health Questionnaire | Evaluated at Baseline and Final (52 days apart) with questions designed to capture function from the prior 4 weeks.
  Self-assessment of functional measures of gastrointestinal health, including colon and small intestinal pain, gastric function, and gastrointestinal inflammation.
Bowel Movement Diary | 52 days
  Daily recording of the number and type (based on Bristol Stool chart) of bowel movements.
Quality of Life Assessment | Evaluated at Baseline and Final (52 days apart)
  Questionnaire that evaluates the impact of gastrointestinal health on daily activities as well as social and psychological impacts.

SECONDARY OUTCOMES:
Gut microbiota changes (beta-diversity) | 2 samples per person, collected ~7 weeks apart
  16s amplicon sequencing of stool samples will be conducted and analyzed for beta-diversity (differences between samples) using principle coordinate analysis of Bray Curtis distances.
Gut microbiota changes (alpha diversity) | 2 samples per person, collected ~7 weeks apart
  16s amplicon sequencing of stool samples will be conducted and analyzed for alpha diversity differences by applying actual and boot-strapped species number estimates, and Shannon and Simpson diversity indices.
Intestinal inflammation | 2 samples per person, collected ~7 weeks apart
  Intestinal inflammation will be assessed by levels of fecal calprotectin measured by ELISA
Intestinal inflammation | 2 samples per person, collected ~7 weeks apart
  Intestinal inflammation will be assessed by levels of secretory immunoglobin A measured by ELISA
Systemic inflammation | 2 blood samples per person, collected ~7 weeks apart
  Human T-cell associated markers of inflammation in the blood will be measured using a multi-plex Luminex panel for 13 analytes.
Systemic inflammation | 2 blood samples per person, collected ~7 weeks apart
  Cultured PBMCs will be stimulated with bacterial LPS and the supernatants will be analyzed for TNF-alpha, Il-6, 1l-10 and IFN-gamma using ELISA.
Lipid panels | 2 blood samples per person, collected ~7 weeks apart
  The Piccolo Xpress lipid panel will be used with a 200ul blood sample to measure total cholesterol and other blood lipid parameters.

OTHER OUTCOMES:
Body Weight | Evaluated at baseline and final visits (~52 days)
  At baseline and final visits, body weight will be measured and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany L Weir, MSc,PhD, Principal Investigator — Colorado State University
Locations (1):
- Food and Nutrition Clinical Research Lab(FNCRL), Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freedman KE, Hill JL, Wei Y, Vazquez AR, Grubb DS, Trotter RE, Wrigley SD, Johnson SA, Foster MT, Weir TL. Examining the Gastrointestinal and Immunomodulatory Effects of the Novel Probiotic Bacillus subtilis DE111. Int J Mol Sci. 2021 Feb 28;22(5):2453. doi: 10.3390/ijms22052453. PMID 33671071
- [Background] Grubb DS, Wrigley SD, Freedman KE, Wei Y, Vazquez AR, Trotter RE, Wallace TC, Johnson SA, Weir TL. PHAGE-2 Study: Supplemental Bacteriophages Extend Bifidobacterium animalis subsp. lactis BL04 Benefits on Gut Health and Microbiota in Healthy Adults. Nutrients. 2020 Aug 17;12(8):2474. doi: 10.3390/nu12082474. PMID 32824480
- [Background] Trotter RE, Vazquez AR, Grubb DS, Freedman KE, Grabos LE, Jones S, Gentile CL, Melby CL, Johnson SA, Weir TL. Bacillus subtilis DE111 intake may improve blood lipids and endothelial function in healthy adults. Benef Microbes. 2020 Nov 15;11(7):621-630. doi: 10.3920/BM2020.0039. Epub 2020 Nov 9. PMID 33161737
- [Background] Gindin M, Febvre HP, Rao S, Wallace TC, Weir TL. Bacteriophage for Gastrointestinal Health (PHAGE) Study: Evaluating the Safety and Tolerability of Supplemental Bacteriophage Consumption. J Am Coll Nutr. 2019 Jan;38(1):68-75. doi: 10.1080/07315724.2018.1483783. Epub 2018 Aug 29. PMID 30157383
- [Background] Febvre HP, Rao S, Gindin M, Goodwin NDM, Finer E, Vivanco JS, Lu S, Manter DK, Wallace TC, Weir TL. PHAGE Study: Effects of Supplemental Bacteriophage Intake on Inflammation and Gut Microbiota in Healthy Adults. Nutrients. 2019 Mar 20;11(3):666. doi: 10.3390/nu11030666. PMID 30897686
- See also: Commercial website for phage product used in the study — https://www.preforpro.com/